CLINICAL TRIAL: NCT01229865
Title: Safety and Efficacy of VB-111 in Subjects With Advanced Differentiated Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vascular Biogenics Ltd. operating as VBL Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VB-111-103
Record Dates: First submitted 2010-10-26; First posted 2010-10-28 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2015-03

CONDITIONS: Differential Thyroid Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VB-111 (Experimental): antiangiogenic and vascular disruptive agent
  Interventions: Drug: VB-111

INTERVENTIONS:
Drug: VB-111

SUMMARY:
The purpose of this study is to examine the safety and evaluate the response of VB-111 on DTC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced DTC (papillary, follicular, Hurthle cell);
2. Absence of sensitivity to therapeutic radioiodine;
3. Measurable disease, defined as at least one non-bony lesion that can be accurately measured in at least one dimension as confirmed with spiral CT scan
4. Life expectancy >3 months; ECOG performance status (PS) 0, 1, or 2; Karnofsky performance status of ≥60%;
5. Subjects with a normal/acceptable hematological profile
6. Subjects with adequate renal function

Exclusion Criteria:

1. Presence of any of the following:

   * Radiotherapy or chemotherapy <4 weeks prior to baseline visit; (Concurrent and/or prior therapy with octreotide will be allowed, provided tumor progression on this therapy has been demonstrated; Concurrent and/or prior therapy with biphosphonates will be allowed)
   * Radiotherapy to ≥25% of bone marrow;
2. Major surgery <4 weeks prior to baseline visit;
3. Any other ongoing investigational agents within 4 weeks before dosing;
4. Subjects who suffered from an acute cardiac event within the last 12 months, including myocardial infarction, cardiac arrythmia, admission for unstable angina, cardiac angioplasty, or stenting;
5. QTc prolongation (defined as QTc interval ≥500 msecs) or other significant ECG abnormalities (e.g. frequent ventricular ectopy, evidence of ongoing myocardial ischemia);
6. Subjects with active vascular disease, either myocardial or peripheral;
7. Subjects with proliferative and/or vascular retinopathy;
8. Subjects with known active liver disease (alcoholic, drug/toxin induced, genetic, or autoimmune) other than related to tumor metastases;
9. Subjects with known CNS metastatic disease (Exception: Subjects with treated CNS metastases stable by radiographic examinations >6 months after definitive therapy administered, are eligible);
10. Subjects testing positive to one of the following viruses: HIV, HBV or HCV;
11. Any of the following conditions:

    * Serious or non-healing wound, ulcer, or bone fracture;
    * History of abdominal fistula, gastro-intestinal perforation, active diverticulitis, intra-abdominal abscess or gastro-intestinal tract bleeding within 6 months of dosing;
    * Any history of cerebrovascular accident (CVA) within 6 months of dosing;
    * Current use of therapeutic warfarin (Note: Low molecular weight heparin and prophylactic low-dose warfarin [INR<1.2 X ULN] are permitted);
    * History of bleeding disorder, including subjects with hemophilia, disseminated intravascular coagulation (DIC), or any other abnormality of coagulation potentially predisposing subjects to bleeding;
    * Poorly controlled depression or anxiety disorder, or recent (within the previous 6 months) suicidal ideation;
12. Subjects with an ongoing requirement for immunosuppressive treatment, including the use of glucocorticoids or cyclosporin, or with a history of chronic use of any such medication within the last 4 weeks before dosing;
13. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-12; Primary Completion 2014-10 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 6 months
Objective response | 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mayo Clinic, Jacksonville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota